CLINICAL TRIAL: NCT03394755
Title: A Phase I, Multi-Center, Open-Label, Dose Escalation Study of Thrombosomes® in Bleeding Thrombocytopenic Patients in Three Cohorts
Brief Title: Thrombosomes® in Bleeding Thrombocytopenic Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cellphire Therapeutics, Inc. (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2017-1
Record Dates: First submitted 2018-01-03; First posted 2018-01-09 (Actual); Results first posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Thrombocytopenia; Hematologic Diseases; Bone Marrow Aplasia
Keywords: thrombocytopenia; bleeding
MeSH Terms: conditions — Thrombocytopenia; Hematologic Diseases; Anemia, Aplastic; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 9.45 x 10^7 Thrombosomes/kg (Experimental): Cohort 1
  Interventions: Biological: Thrombosomes
- 1.89 x 10^8 Thrombosomes/kg (Experimental): Cohort 2
  Interventions: Biological: Thrombosomes
- 3.78 x10^8 Thrombosomes/kg (Experimental): Cohort 3
  Interventions: Biological: Thrombosomes

INTERVENTIONS:
Biological: Thrombosomes — Freeze-dried platelets

SUMMARY:
The study evaluates the safety and potential early signals of efficacy of allogeneic Thrombosomes in bleeding thrombocytopenic patients

DETAILED DESCRIPTION:
The primary objective of the present study was to assess the safety of increasing dose levels of Thrombosomes in bleeding patients with thrombocytopenia. The secondary objective was to explore early signals of clinical efficacy of Thrombosomes in this population. The secondary objectives included: 1) Evaluation of the impact on WHO (World Health Organization) bleeding scores at various timepoints; 2) number and type of blood products infused through day 6 follow-up period; and 3) post hoc analysis of hematology, coagulation, and chemistry.

ELIGIBILITY:
Inclusion Criteria:

* Adults up to 74 y/o with any of following: acute leukemia (ALL or AML), myelodysplasia, aplasia, and/or therapy (chemotherapy or radiation) induced bone marrow aplasia or hypoplasia with thrombocytopenia (platelet count ≥ 5,000 and ≤ 70,000/μL) for a minimum of 2 days. May include bone marrow transplant or peripheral or cord blood stem cell recipients, but not subjects with Graft-vs-Host disease.
* Hospitalized patients (or willing to be hospitalized for 24 hours after Rx) with Modified WHO Grade 1 (subset) or Grade 2 Bleeding Score or at risk for same within 4 weeks of screening. The Grade 1 subset includes patients who have either epistaxis, hematuria, oral petechiae, or bleeding at invasive or other wound sites.
* No platelet inhibitor drugs within 5 days prior to infusion and through Day 6 follow-up period.

Exclusion Criteria:

* History or condition related to thrombosis, embolism or vascular occlusion/ischemia, including but not limited to: transient ischemic attack, stroke, myocardial infarction, stent placement, valve replacement and/or repair
* Currently with an active acute infection, or suspected infection, a single oral temperature of ≥ 101° F or a temperature of ≥ 100.4°F sustained over a 1 h period in past 24 h. Subjects on prophylactic antibiotics are not excluded from study
* Coagulopathy or receiving anticoagulants that result in PT (prothrombin time) or aPTT (activated partial thromboplastin time) values greater than 1.3 X upper limit of normal or elevated D-dimer of decreased fibrinogen
* History of any inherited coagulation or platelet function, disorder or ITP (idiopathic thrombocytopenic purpura), TTP (thrombotic thrombocytopenic purpura), or HUS (hemolytic-uremic syndrome)
* Receipt of tranexamic acid or other antifibrinolytics within 48 hrs prior to infusion
* Treatment with an investigational drug within 1 month of infusion, other than for treatment of their underlying disease

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fitzpatrick, Study Director — Cellphire Therapeutics, Inc.
Locations (7):
- United States (6):
  - City of Hope, Duarte, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Michigan, Ann Arbor, Michigan
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hoxworth Blood Center/University of Cincinnati, Cincinnati, Ohio
  - MD Anderson Cancer Center, Houston, Texas
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ohanian M, Cancelas JA, Davenport R, Pullarkat V, Hervig T, Broome C, Marek K, Kelly M, Gul Z, Rugg N, Nestheide S, Kinne B, Szczepiorkowski Z, Kantarjian H, Pehta J, Biehl R, Yu A, Aung F, Antebi B, Fitzpatrick GM. Freeze-dried platelets are a promising alternative in bleeding thrombocytopenic patients with hematological malignancies. Am J Hematol. 2022 Mar 1;97(3):256-266. doi: 10.1002/ajh.26403. Epub 2021 Dec 23. PMID 34748664

RESULTS

PARTICIPANT FLOW:
Groups:
- 9.45 x 10^7 Thrombosomes/kg: Cohort 1: Thrombosomes: Freeze-dried platelets
- 1.89 x 10^8 Thrombosomes/kg: Cohort 2: Thrombosomes: Freeze-dried platelets
- 3.78 x 10^8 Thrombosomes/kg: Cohort 3: Thrombosomes: Freeze-dried platelets
Period: Overall Study
Arm/Group | 9.45 x 10^7 Thrombosomes/kg | 1.89 x 10^8 Thrombosomes/kg | 3.78 x 10^8 Thrombosomes/kg
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Thrombosomes 94.5 Million Particles/kg Body Weight; Thrombosomes 189 Million Particles/kg Body Weight; 378 Million Particles/kg Body Weight: Thrombosomes: Freeze-dried platelet derived hemostatic
- Total: Total of all reporting groups
Arm/Group | Thrombosomes 94.5 Million Particles/kg Body Weight | Thrombosomes 189 Million Particles/kg Body Weight | 378 Million Particles/kg Body Weight | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Continuous [Median (Full Range); unit: years] | 55.5 [27 to 63] | 59.5 [24 to 66] | 60.5 [26 to 71] | 59 [24 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 3 | 10
  Male | 5 | 4 | 5 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 8 | 6 | 7 | 21
  Unknown or Not Reported | 0 | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 3 | 4
  White | 7 | 7 | 4 | 18
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2
Safety Population [Count of Participants; unit: Participants] | 8 | 8 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Treatment-Emergent Adverse Events (TEAE)
Description: Overall frequency of (and number and percentage of patients who experience) TEAEs including serious adverse drug reactions and treatment-related events specifically defining the study's suspension and stopping rules (i.e., thromboembolic events, acute lung injury, anaphylaxis, and death).
Time Frame: 30 days
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- Thrombosomes 378 Million Particles/kg Body Weight: Thrombosomes: Freeze-dried platelet derived hemostatic
Arm/Group | Thrombosomes 94.5 Million Particles/kg Body Weight | Thrombosomes 189 Million Particles/kg Body Weight | Thrombosomes 378 Million Particles/kg Body Weight
Number analyzed (Participants) | 8 | 8 | 8
Participants | 7 | 6 | 5

2. Primary Outcome: Number of Patients With Treatment-Emergent Serious Adverse Events (TESAE)
Description: Overall frequency of (and number and percentage of patients who experience) TESAEs including serious adverse drug reactions and treatment-related events specifically defining the study's suspension and stopping rules (i.e., thromboembolic events, acute lung injury, anaphylaxis, and death).
Time Frame: 30 days
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Thrombosomes 94.5 Million Particles/kg Body Weight | Thrombosomes 189 Million Particles/kg Body Weight | Thrombosomes 378 Million Particles/kg Body Weight
Number analyzed (Participants) | 8 | 8 | 8
Participants | 1 | 5 | 4

3. Secondary Outcome: Number of WHO Bleeding Sites With Status Change From Baseline
Description: Grade-level change in WHO bleeding assessment score at most severe bleeding site from baseline; WHO bleeding assessment score ranges from 1 to 4, with higher numbers indicating worse bleeding.
Time Frame: 1, 6, 24 hours, and Day 6 post infusion
Population: All bleeding sites among the evaluable patient population were grouped into a change in WHO bleeding status rather than by treatment arms.
Measure: Count of Units; unit: Total bleeding sites
Units Other Than Participants: Total bleeding sites
Groups:
- Worsened; No Change; Improved: Bleeding sites post infusion
Arm/Group | Worsened | No Change | Improved
Number analyzed (Participants) | 22 | 22 | 22
Number analyzed (Total bleeding sites) | 27 | 27 | 27
Total bleeding sites
  1 hour post infusion | 0 | 24 | 3
  6hrs post infusion | 0 | 21 | 6
  24 hours post infusion | 0 | 17 | 10
  Day 6 | 0 | 10 | 17

4. Secondary Outcome: Number of Patients With Grade-level Change in WHO Bleeding Assessment Score From Baseline - Patients WHO Score at Primary Bleeding Site
Description: Patients WHO score at primary bleeding site. WHO bleeding assessment score ranges from 1 to 4, with higher numbers indicating worse bleeding. The maximum WHO bleeding assessment score for patients on study was 2.
Time Frame: Baseline, 1, 6, 24 hours, and Day 6 post infusion
Population: The evaluable patient population is grouped by WHO grade levels 0, 1, and 2 rather than by treatment arms.
Measure: Count of Participants; unit: Participants
Groups:
- Grade 0; Grade 1; Grade 2: Grade at bleeding site post infusion
Arm/Group | Grade 0 | Grade 1 | Grade 2
Number analyzed (Participants) | 22 | 22 | 22
Participants
  Baseline | 0 | 7 | 15
  1 hour post infusion | 1 | 7 | 14
  6 hours post infusion | 3 | 7 | 12
  24 hours post infusion | 4 | 6 | 12
  Day 6 | 8 | 6 | 8

5. Secondary Outcome: Number of Patients With a Shift From Baseline in Hemoglobin
Description: Shift from baseline clinical status of hemoglobin measure at different timepoints post infusion
Time Frame: 1, 6, 24 hours, Day 3, 4, 5, and 6 post infusion
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Thrombosomes 94.5 Million Particles/kg Body Weight | Thrombosomes 189 Million Particles/kg Body Weight | Thrombosomes 378 Million Particles/kg Body Weight
Number analyzed (Participants) | 8 | 8 | 8
Participants
  1 hour post infusion: number analyzed (Participants) | 7 | 8 | 7
  1 hour post infusion: Normal>Normal | 0 | 0 | 0
  1 hour post infusion: Normal>Abnormal Not Clinically Significant | 0 | 0 | 0
  1 hour post infusion: Normal>Abnormal Clinically Significant | 0 | 0 | 0
  1 hour post infusion: Abnormal Not Clinically Significant> Normal | 0 | 0 | 0
  1 hour post infusion: Abnormal Not Clinically Significant>Abnormal Not Clinically Significant | 6 | 7 | 7
  1 hour post infusion: Abnormal Not Clinically Significant>Abnormal Clinically Significant | 0 | 0 | 0
  1 hour post infusion: Abnormal Clinically Significant>Normal | 0 | 0 | 0
  1 hour post infusion: Abnormal Clinically Significant>Abnormal Not Clinically Significant | 0 | 0 | 0
  1 hour post infusion: Abnormal Clinically Significant>Abnormal Clinically Significant | 1 | 1 | 0
  6 hours post infusion: number analyzed (Participants) | 6 | 8 | 7
  6 hours post infusion: Normal>Normal | 0 | 0 | 0
  6 hours post infusion: Normal>Abnormal Not Clinically Significant | 0 | 0 | 0
  6 hours post infusion: Normal>Abnormal Clinically Significant | 0 | 0 | 0
  6 hours post infusion: Abnormal Not Clinically Significant> Normal | 0 | 0 | 0
  6 hours post infusion: Abnormal Not Clinically Significant>Abnormal Not Clinically Significant | 4 | 7 | 7
  6 hours post infusion: Abnormal Not Clinically Significant>Abnormal Clinically Significant | 1 | 0 | 0
  6 hours post infusion: Abnormal Clinically Significant>Normal | 0 | 0 | 0
  6 hours post infusion: Abnormal Clinically Significant>Abnormal Not Clinically Significant | 0 | 0 | 0
  6 hours post infusion: Abnormal Clinically Significant>Abnormal Clinically Significant | 1 | 1 | 0
  24 hours post infusion: Normal>Normal | 0 | 0 | 0
  24 hours post infusion: Normal>Abnormal Not Clinically Significant | 0 | 0 | 0
  24 hours post infusion: Normal>Abnormal Clinically Significant | 0 | 0 | 0
  24 hours post infusion: Abnormal Not Clinically Significant> Normal | 0 | 0 | 0
  24 hours post infusion: Abnormal Not Clinically Significant>Abnormal Not Clinically Significant | 7 | 7 | 8
  24 hours post infusion: Abnormal Not Clinically Significant>Abnormal Clinically Significant | 0 | 0 | 0
  24 hours post infusion: Abnormal Clinically Significant>Normal | 0 | 0 | 0
  24 hours post infusion: Abnormal Clinically Significant>Abnormal Not Clinically Significant | 0 | 1 | 0
  24 hours post infusion: Abnormal Clinically Significant>Abnormal Clinically Significant | 1 | 0 | 0
  Day 3: number analyzed (Participants) | 8 | 8 | 6
  Day 3: Normal>Normal | 0 | 0 | 0
  Day 3: Normal>Abnormal Not Clinically Significant | 0 | 0 | 0
  Day 3: Normal>Abnormal Clinically Significant | 0 | 0 | 0
  Day 3: Abnormal Not Clinically Significant> Normal | 0 | 0 | 0
  Day 3: Abnormal Not Clinically Significant>Abnormal Not Clinically Significant | 6 | 7 | 6
  Day 3: Abnormal Not Clinically Significant>Abnormal Clinically Significant | 1 | 0 | 0
  Day 3: Abnormal Clinically Significant>Normal | 0 | 0 | 0
  Day 3: Abnormal Clinically Significant>Abnormal Not Clinically Significant | 1 | 1 | 0
  Day 3: Abnormal Clinically Significant>Abnormal Clinically Significant | 0 | 0 | 0
  Day 4: number analyzed (Participants) | 7 | 8 | 5
  Day 4: Normal>Normal | 0 | 0 | 0
  Day 4: Normal>Abnormal Not Clinically Significant | 0 | 0 | 0
  Day 4: Normal>Abnormal Clinically Significant | 0 | 0 | 0
  Day 4: Abnormal Not Clinically Significant> Normal | 0 | 0 | 0
  Day 4: Abnormal Not Clinically Significant>Abnormal Not Clinically Significant | 4 | 7 | 5
  Day 4: Abnormal Not Clinically Significant>Abnormal Clinically Significant | 2 | 0 | 0
  Day 4: Abnormal Clinically Significant>Normal | 0 | 0 | 0
  Day 4: Abnormal Clinically Significant>Abnormal Not Clinically Significant | 1 | 1 | 0
  Day 4: Abnormal Clinically Significant>Abnormal Clinically Significant | 0 | 0 | 0
  Day 5: number analyzed (Participants) | 7 | 8 | 5
  Day 5: Normal>Normal | 0 | 0 | 0
  Day 5: Normal>Abnormal Not Clinically Significant | 0 | 0 | 0
  Day 5: Normal>Abnormal Clinically Significant | 0 | 0 | 0
  Day 5: Abnormal Not Clinically Significant> Normal | 0 | 0 | 0
  Day 5: Abnormal Not Clinically Significant>Abnormal Not Clinically Significant | 5 | 7 | 5
  Day 5: Abnormal Not Clinically Significant>Abnormal Clinically Significant | 1 | 0 | 0
  Day 5: Abnormal Clinically Significant>Normal | 0 | 0 | 0
  Day 5: Abnormal Clinically Significant>Abnormal Not Clinically Significant | 1 | 0 | 0
  Day 5: Abnormal Clinically Significant>Abnormal Clinically Significant | 0 | 1 | 0
  Day 6: Normal>Normal | 0 | 0 | 0
  Day 6: Normal>Abnormal Not Clinically Significant | 0 | 0 | 0
  Day 6: Normal>Abnormal Clinically Significant | 0 | 0 | 0
  Day 6: Abnormal Not Clinically Significant> Normal | 0 | 0 | 0
  Day 6: Abnormal Not Clinically Significant>Abnormal Not Clinically Significant | 5 | 7 | 8
  Day 6: Abnormal Not Clinically Significant>Abnormal Clinically Significant | 2 | 0 | 0
  Day 6: Abnormal Clinically Significant>Normal | 0 | 0 | 0
  Day 6: Abnormal Clinically Significant>Abnormal Not Clinically Significant | 1 | 1 | 0
  Day 6: Abnormal Clinically Significant>Abnormal Clinically Significant | 0 | 0 | 0

6. Secondary Outcome: Number of Patients With a Shift From Baseline in Hematocrit
Description: Shift from baseline clinical status of hematocrit measure at different timepoints post infusion
Time Frame: 1, 6, 24 hours, Day 3, 4, 5, and 6 post infusion
Population: Safety population with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Thrombosomes 94.5 Million Particles/kg Body Weight | Thrombosomes 189 Million Particles/kg Body Weight | Thrombosomes 378 Million Particles/kg Body Weight
Number analyzed (Participants) | 8 | 8 | 8
Participants
  1 hour post infusion: number analyzed (Participants) | 7 | 8 | 7
  1 hour post infusion: Normal>Normal | 0 | 0 | 0
  1 hour post infusion: Normal>Abnormal NCS | 0 | 0 | 0
  1 hour post infusion: Normal>Abnormal CS | 0 | 0 | 0
  1 hour post infusion: Abnormal NCS> Normal | 0 | 0 | 0
  1 hour post infusion: Abnormal NCS>Abnormal NCS | 7 | 7 | 7
  1 hour post infusion: Abnormal NCS>Abnormal CS | 0 | 0 | 0
  1 hour post infusion: Abnormal CS>Normal | 0 | 0 | 0
  1 hour post infusion: Abnormal CS>Abnormal NCS | 0 | 0 | 0
  1 hour post infusion: Abnormal CS>Abnormal CS | 0 | 1 | 0
  6 hours post infusion: number analyzed (Participants) | 6 | 8 | 8
  6 hours post infusion: Normal>Normal | 0 | 0 | 0
  6 hours post infusion: Normal>Abnormal NCS | 0 | 0 | 0
  6 hours post infusion: Normal>Abnormal CS | 0 | 0 | 0
  6 hours post infusion: Abnormal NCS> Normal | 0 | 0 | 0
  6 hours post infusion: Abnormal NCS>Abnormal NCS | 5 | 7 | 8
  6 hours post infusion: Abnormal NCS>Abnormal CS | 1 | 0 | 0
  6 hours post infusion: Abnormal CS>Normal | 0 | 0 | 0
  6 hours post infusion: Abnormal CS>Abnormal NCS | 0 | 1 | 0
  6 hours post infusion: Abnormal CS>Abnormal CS | 0 | 0 | 0
  24 hours post infusion: Normal>Normal | 0 | 0 | 0
  24 hours post infusion: Normal>Abnormal NCS | 0 | 0 | 0
  24 hours post infusion: Normal>Abnormal CS | 0 | 0 | 0
  24 hours post infusion: Abnormal NCS> Normal | 0 | 0 | 0
  24 hours post infusion: Abnormal NCS>Abnormal NCS | 7 | 7 | 8
  24 hours post infusion: Abnormal NCS>Abnormal CS | 0 | 0 | 0
  24 hours post infusion: Abnormal CS>Normal | 0 | 0 | 0
  24 hours post infusion: Abnormal CS>Abnormal NCS | 1 | 1 | 0
  24 hours post infusion: Abnormal CS>Abnormal CS | 0 | 0 | 0
  Day 3: number analyzed (Participants) | 8 | 8 | 6
  Day 3: Normal>Normal | 0 | 0 | 0
  Day 3: Normal>Abnormal NCS | 0 | 0 | 0
  Day 3: Normal>Abnormal CS | 0 | 0 | 0
  Day 3: Abnormal NCS> Normal | 0 | 0 | 0
  Day 3: Abnormal NCS>Abnormal NCS | 7 | 7 | 6
  Day 3: Abnormal NCS>Abnormal CS | 0 | 0 | 0
  Day 3: Abnormal CS>Normal | 0 | 0 | 0
  Day 3: Abnormal CS>Abnormal NCS | 1 | 1 | 0
  Day 3: Abnormal CS>Abnormal CS | 0 | 0 | 0
  Day 4: number analyzed (Participants) | 7 | 8 | 5
  Day 4: Normal>Normal | 0 | 0 | 0
  Day 4: Normal>Abnormal NCS | 0 | 0 | 0
  Day 4: Normal>Abnormal CS | 0 | 0 | 0
  Day 4: Abnormal NCS> Normal | 0 | 0 | 0
  Day 4: Abnormal NCS>Abnormal NCS | 6 | 7 | 5
  Day 4: Abnormal NCS>Abnormal CS | 1 | 0 | 0
  Day 4: Abnormal CS>Normal | 0 | 0 | 0
  Day 4: Abnormal CS>Abnormal NCS | 0 | 1 | 0
  Day 4: Abnormal CS>Abnormal CS | 0 | 0 | 0
  Day 5: number analyzed (Participants) | 7 | 8 | 5
  Day 5: Normal>Normal | 0 | 0 | 0
  Day 5: Normal>Abnormal NCS | 0 | 0 | 0
  Day 5: Normal>Abnormal CS | 0 | 0 | 0
  Day 5: Abnormal NCS> Normal | 0 | 0 | 0
  Day 5: Abnormal NCS>Abnormal NCS | 7 | 7 | 5
  Day 5: Abnormal NCS>Abnormal CS | 0 | 0 | 0
  Day 5: Abnormal CS>Normal | 0 | 0 | 0
  Day 5: Abnormal CS>Abnormal NCS | 0 | 0 | 0
  Day 5: Abnormal CS>Abnormal CS | 0 | 1 | 0
  Day 6: Normal>Normal | 0 | 0 | 0
  Day 6: Normal>Abnormal NCS | 0 | 0 | 0
  Day 6: Normal>Abnormal CS | 0 | 0 | 0
  Day 6: Abnormal NCS> Normal | 0 | 0 | 0
  Day 6: Abnormal NCS>Abnormal NCS | 6 | 7 | 8
  Day 6: Abnormal NCS>Abnormal CS | 1 | 0 | 0
  Day 6: Abnormal CS>Normal | 0 | 0 | 0
  Day 6: Abnormal CS>Abnormal NCS | 1 | 1 | 0
  Day 6: Abnormal CS>Abnormal CS | 0 | 0 | 0

7. Secondary Outcome: Number or Patients With a Shift From Baseline in Coagulation Measures 24 Hours Post Infusion
Description: Shift from baseline clinical status of coagulation measure at 24 hours post infusion for each cohort
Time Frame: 24 hours post infusion
Population: Safety population with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Thrombosomes 94.5 Million Particles/kg Body Weight | Thrombosomes 189 Million Particles/kg Body Weight | Thrombosomes 378 Million Particles/kg Body Weight
Number analyzed (Participants) | 8 | 8 | 8
Participants
  Prothrombin Time (PT): number analyzed (Participants) | 8 | 7 | 7
  Prothrombin Time (PT): Normal>Normal | 6 | 5 | 5
  Prothrombin Time (PT): Normal>Abnormal Not Clinically Significant | 0 | 1 | 0
  Prothrombin Time (PT): Normal>Abnormal Clinically Significant | 0 | 0 | 0
  Prothrombin Time (PT): Abnormal Not Clinically Significant> Normal | 0 | 0 | 1
  Prothrombin Time (PT): Abnormal Not Clinically Significant>Abnormal Not Clinically Significant | 2 | 1 | 1
  Prothrombin Time (PT): Abnormal Not Clinically Significant>Abnormal Clinically Significant | 0 | 0 | 0
  Prothrombin Time (PT): Abnormal Clinically Significant>Normal | 0 | 0 | 0
  Prothrombin Time (PT): Abnormal Clinically Significant>Abnormal Not Clinically Significant | 0 | 0 | 0
  Prothrombin Time (PT): Abnormal Clinically Significant>Abnormal Clinically Significant | 0 | 0 | 0
  International Normalized Ratio (INR): number analyzed (Participants) | 8 | 8 | 7
  International Normalized Ratio (INR): Normal>Normal | 7 | 7 | 6
  International Normalized Ratio (INR): Normal>Abnormal Not Clinically Significant | 0 | 1 | 0
  International Normalized Ratio (INR): Normal>Abnormal Clinically Significant | 0 | 0 | 0
  International Normalized Ratio (INR): Abnormal Not Clinically Significant> Normal | 0 | 0 | 1
  International Normalized Ratio (INR): Abnormal Not Clinically Significant>Abnormal Not Clinically Significant | 1 | 0 | 0
  International Normalized Ratio (INR): Abnormal Not Clinically Significant>Abnormal Clinically Significant | 0 | 0 | 0
  International Normalized Ratio (INR): Abnormal Clinically Significant>Normal | 0 | 0 | 0
  International Normalized Ratio (INR): Abnormal Clinically Significant>Abnormal Not Clinically Significant | 0 | 0 | 0
  International Normalized Ratio (INR): Abnormal Clinically Significant>Abnormal Clinically Significant | 0 | 0 | 0
  Activated Partial Thromboplastin Time (aPTT): number analyzed (Participants) | 7 | 8 | 6
  Activated Partial Thromboplastin Time (aPTT): Normal>Normal | 2 | 6 | 4
  Activated Partial Thromboplastin Time (aPTT): Normal>Abnormal Not Clinically Significant | 1 | 0 | 0
  Activated Partial Thromboplastin Time (aPTT): Normal>Abnormal Clinically Significant | 0 | 0 | 0
  Activated Partial Thromboplastin Time (aPTT): Abnormal Not Clinically Significant> Normal | 1 | 0 | 1
  Activated Partial Thromboplastin Time (aPTT): Abnormal Not Clinically Significant>Abnormal Not Clinically Significant | 3 | 2 | 1
  Activated Partial Thromboplastin Time (aPTT): Abnormal Not Clinically Significant>Abnormal Clinically Significant | 0 | 0 | 0
  Activated Partial Thromboplastin Time (aPTT): Abnormal Clinically Significant>Normal | 0 | 0 | 0
  Activated Partial Thromboplastin Time (aPTT): Abnormal Clinically Significant>Abnormal Not Clinically Significant | 0 | 0 | 0
  Activated Partial Thromboplastin Time (aPTT): Abnormal Clinically Significant>Abnormal Clinically Significant | 0 | 0 | 0
  D-dimer: number analyzed (Participants) | 7 | 8 | 7
  D-dimer: Normal>Normal | 0 | 0 | 0
  D-dimer: Normal>Abnormal Not Clinically Significant | 0 | 0 | 1
  D-dimer: Normal>Abnormal Clinically Significant | 0 | 0 | 0
  D-dimer: Abnormal Not Clinically Significant> Normal | 0 | 1 | 0
  D-dimer: Abnormal Not Clinically Significant>Abnormal Not Clinically Significant | 6 | 7 | 6
  D-dimer: Abnormal Not Clinically Significant>Abnormal Clinically Significant | 0 | 0 | 0
  D-dimer: Abnormal Clinically Significant>Normal | 0 | 0 | 0
  D-dimer: Abnormal Clinically Significant>Abnormal Not Clinically Significant | 0 | 0 | 0
  D-dimer: Abnormal Clinically Significant>Abnormal Clinically Significant | 1 | 0 | 0
  Fibrinogen: number analyzed (Participants) | 7 | 8 | 7
  Fibrinogen: Normal>Normal | 2 | 5 | 3
  Fibrinogen: Normal>Abnormal Not Clinically Significant | 1 | 0 | 0
  Fibrinogen: Normal>Abnormal Clinically Significant | 0 | 0 | 0
  Fibrinogen: Abnormal Not Clinically Significant> Normal | 0 | 0 | 1
  Fibrinogen: Abnormal Not Clinically Significant>Abnormal Not Clinically Significant | 4 | 3 | 3
  Fibrinogen: Abnormal Not Clinically Significant>Abnormal Clinically Significant | 0 | 0 | 0
  Fibrinogen: Abnormal Clinically Significant>Normal | 0 | 0 | 0
  Fibrinogen: Abnormal Clinically Significant>Abnormal Not Clinically Significant | 0 | 0 | 0
  Fibrinogen: Abnormal Clinically Significant>Abnormal Clinically Significant | 0 | 0 | 0
  Thrombin Antithrombin (TAT): Normal>Normal | 1 | 2 | 2
  Thrombin Antithrombin (TAT): Normal>Abnormal Not Clinically Significant | 0 | 1 | 1
  Thrombin Antithrombin (TAT): Normal>Abnormal Clinically Significant | 0 | 0 | 0
  Thrombin Antithrombin (TAT): Abnormal Not Clinically Significant> Normal | 1 | 1 | 0
  Thrombin Antithrombin (TAT): Abnormal Not Clinically Significant>Abnormal Not Clinically Significant | 4 | 4 | 5
  Thrombin Antithrombin (TAT): Abnormal Not Clinically Significant>Abnormal Clinically Significant | 0 | 0 | 0
  Thrombin Antithrombin (TAT): Abnormal Clinically Significant>Normal | 0 | 0 | 0
  Thrombin Antithrombin (TAT): Abnormal Clinically Significant>Abnormal Not Clinically Significant | 0 | 0 | 0
  Thrombin Antithrombin (TAT): Abnormal Clinically Significant>Abnormal Clinically Significant | 2 | 0 | 0
  Prothrombin Fragment (PF) 1+2: number analyzed (Participants) | 8 | 7 | 8
  Prothrombin Fragment (PF) 1+2: Normal>Normal | 1 | 2 | 1
  Prothrombin Fragment (PF) 1+2: Normal>Abnormal Not Clinically Significant | 0 | 1 | 0
  Prothrombin Fragment (PF) 1+2: Normal>Abnormal Clinically Significant | 0 | 0 | 0
  Prothrombin Fragment (PF) 1+2: Abnormal Not Clinically Significant> Normal | 0 | 0 | 3
  Prothrombin Fragment (PF) 1+2: Abnormal Not Clinically Significant>Abnormal Not Clinically Significant | 3 | 4 | 4
  Prothrombin Fragment (PF) 1+2: Abnormal Not Clinically Significant>Abnormal Clinically Significant | 1 | 0 | 0
  Prothrombin Fragment (PF) 1+2: Abnormal Clinically Significant>Normal | 0 | 0 | 0
  Prothrombin Fragment (PF) 1+2: Abnormal Clinically Significant>Abnormal Not Clinically Significant | 1 | 0 | 0
  Prothrombin Fragment (PF) 1+2: Abnormal Clinically Significant>Abnormal Clinically Significant | 2 | 0 | 0
  Thrombin Generation Assay (TGA) (Lag Time): number analyzed (Participants) | 7 | 7 | 8
  Thrombin Generation Assay (TGA) (Lag Time): Normal>Normal | 7 | 7 | 7
  Thrombin Generation Assay (TGA) (Lag Time): Normal>Abnormal Not Clinically Significant | 0 | 0 | 0
  Thrombin Generation Assay (TGA) (Lag Time): Normal>Abnormal Clinically Significant | 0 | 0 | 0
  Thrombin Generation Assay (TGA) (Lag Time): Abnormal Not Clinically Significant> Normal | 0 | 0 | 0
  Thrombin Generation Assay (TGA) (Lag Time): Abnormal Not Clinically Significant>Abnormal Not Clinically Significant | 0 | 0 | 1
  Thrombin Generation Assay (TGA) (Lag Time): Abnormal Not Clinically Significant>Abnormal Clinically Significant | 0 | 0 | 0
  Thrombin Generation Assay (TGA) (Lag Time): Abnormal Clinically Significant>Normal | 0 | 0 | 0
  Thrombin Generation Assay (TGA) (Lag Time): Abnormal Clinically Significant>Abnormal Not Clinically Significant | 0 | 0 | 0
  Thrombin Generation Assay (TGA) (Lag Time): Abnormal Clinically Significant>Abnormal Clinically Significant | 0 | 0 | 0
  Thrombin Generation Assay (TGA) (Time to Peak): number analyzed (Participants) | 7 | 7 | 8
  Thrombin Generation Assay (TGA) (Time to Peak): Normal>Normal | 7 | 6 | 4
  Thrombin Generation Assay (TGA) (Time to Peak): Normal>Abnormal Not Clinically Significant | 0 | 0 | 1
  Thrombin Generation Assay (TGA) (Time to Peak): Normal>Abnormal Clinically Significant | 0 | 0 | 0
  Thrombin Generation Assay (TGA) (Time to Peak): Abnormal Not Clinically Significant> Normal | 0 | 1 | 0
  Thrombin Generation Assay (TGA) (Time to Peak): Abnormal Not Clinically Significant>Abnormal Not Clinically Significant | 0 | 0 | 3
  Thrombin Generation Assay (TGA) (Time to Peak): Abnormal Not Clinically Significant>Abnormal Clinically Significant | 0 | 0 | 0
  Thrombin Generation Assay (TGA) (Time to Peak): Abnormal Clinically Significant>Normal | 0 | 0 | 0
  Thrombin Generation Assay (TGA) (Time to Peak): Abnormal Clinically Significant>Abnormal Not Clinically Significant | 0 | 0 | 0
  Thrombin Generation Assay (TGA) (Time to Peak): Abnormal Clinically Significant>Abnormal Clinically Significant | 0 | 0 | 0
  Thrombin Generation Assay (TGA) (Thrombin Peak Height): number analyzed (Participants) | 7 | 7 | 8
  Thrombin Generation Assay (TGA) (Thrombin Peak Height): Normal>Normal | 7 | 7 | 7
  Thrombin Generation Assay (TGA) (Thrombin Peak Height): Normal>Abnormal Not Clinically Significant | 0 | 0 | 1
  Thrombin Generation Assay (TGA) (Thrombin Peak Height): Normal>Abnormal Clinically Significant | 0 | 0 | 0
  Thrombin Generation Assay (TGA) (Thrombin Peak Height): Abnormal Not Clinically Significant> Normal | 0 | 0 | 0
  Thrombin Generation Assay (TGA) (Thrombin Peak Height): Abnormal Not Clinically Significant>Abnormal Not Clinically Significant | 0 | 0 | 0
  Thrombin Generation Assay (TGA) (Thrombin Peak Height): Abnormal Not Clinically Significant>Abnormal Clinically Significant | 0 | 0 | 0
  Thrombin Generation Assay (TGA) (Thrombin Peak Height): Abnormal Clinically Significant>Normal | 0 | 0 | 0
  Thrombin Generation Assay (TGA) (Thrombin Peak Height): Abnormal Clinically Significant>Abnormal Not Clinically Significant | 0 | 0 | 0
  Thrombin Generation Assay (TGA) (Thrombin Peak Height): Abnormal Clinically Significant>Abnormal Clinically Significant | 0 | 0 | 0
  Thrombin Generation Assay (TGA) Endogenous Thrombin Potential (ETP): number analyzed (Participants) | 7 | 7 | 8
  Thrombin Generation Assay (TGA) Endogenous Thrombin Potential (ETP): Normal>Normal | 5 | 6 | 6
  Thrombin Generation Assay (TGA) Endogenous Thrombin Potential (ETP): Normal>Abnormal Not Clinically Significant | 1 | 0 | 1
  Thrombin Generation Assay (TGA) Endogenous Thrombin Potential (ETP): Normal>Abnormal Clinically Significant | 0 | 0 | 0
  Thrombin Generation Assay (TGA) Endogenous Thrombin Potential (ETP): Abnormal Not Clinically Significant> Normal | 1 | 1 | 1
  Thrombin Generation Assay (TGA) Endogenous Thrombin Potential (ETP): Abnormal Not Clinically Significant>Abnormal Not Clinically Significant | 0 | 0 | 0
  Thrombin Generation Assay (TGA) Endogenous Thrombin Potential (ETP): Abnormal Not Clinically Significant>Abnormal Clinically Significant | 0 | 0 | 0
  Thrombin Generation Assay (TGA) Endogenous Thrombin Potential (ETP): Abnormal Clinically Significant>Normal | 0 | 0 | 0
  Thrombin Generation Assay (TGA) Endogenous Thrombin Potential (ETP): Abnormal Clinically Significant>Abnormal Not Clinically Significant | 0 | 0 | 0
  Thrombin Generation Assay (TGA) Endogenous Thrombin Potential (ETP): Abnormal Clinically Significant>Abnormal Clinically Significant | 0 | 0 | 0

8. Secondary Outcome: Median Platelet Counts
Description: Median Platelet Counts Per Time Point
Time Frame: Screening, Baseline, 1, 6, 24 hours, Day 3, 4, 5, and 6 post infusion
Population: The median platelet count of the safety patient population is grouped by timepoints(screening, baseline and post infusion 1, 6, 24 hours, Day 3, 4, 5, 6) rather than by treatment arms.
Measure: Median (Full Range); unit: PLT Count (10³/µl)
Groups:
- Platelets: Median Platelet Count
Arm/Group | Platelets
Number analyzed (Participants) | 24
PLT Count (10³/µl)
  Screening | 16 [8 to 48]
  Baseline | 18.5 [2 to 51]
  1 hour post infusion | 13.5 [2 to 46]
  6 hrs post infusion | 14 [1 to 46]
  24 hrs post infusion | 20.5 [2 to 78]
  Day 3 | 22.5 [3 to 83]
  Day 4 | 18.5 [3 to 106]
  Day 5 | 20 [6 to 146]
  Day 6 | 18 [2 to 275]

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) were recorded starting from the day of infusion (Day 1). For non-serious AEs, recording was through the Day 6 visit, and for serious adverse events (SAEs), recording was through the Day 30 visit (phone assessment was acceptable), or until premature discontinuation occurred. AEs were assessed by investigator at visits by physician exam, by vital signs, by laboratory assessments, by chart review, and by open-ended patient query.
Description: Information is reported on treatment-emergent AEs and SAEs (TEAEs and TESAEs).
Arm/Group | Thrombosomes 94.5 Million Particles/kg Body Weight | Thrombosomes 189 Million Particles/kg Body Weight | Thrombosomes 378 Million Particles/kg Body Weight
All-Cause Mortality (participants affected / at risk) | 0/8 | 3/8 | 3/8
Serious Adverse Events (participants affected / at risk) | 1/8 | 5/8 | 4/8
Other Adverse Events (participants affected / at risk) | 7/8 | 6/8 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Thrombosomes 94.5 Million Particles/kg Body Weight (N=8) | Thrombosomes 189 Million Particles/kg Body Weight (N=8) | Thrombosomes 378 Million Particles/kg Body Weight (N=8)
Sepsis (Infections and infestations) | 0 | 1 | 2
Bacteremia (Infections and infestations) | 0 | 1 | 0
Cholecystitis infective (Infections and infestations) | 0 | 1 | 0
Encephalitis viral (Infections and infestations) | 0 | 0 | 1
Pathogen resistance (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1
Necrosis (General disorders) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Pituitary haemorrhage (Endocrine disorders) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Acute graft versus host disease (Immune system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Thrombosomes 94.5 Million Particles/kg Body Weight (N=8) | Thrombosomes 189 Million Particles/kg Body Weight (N=8) | Thrombosomes 378 Million Particles/kg Body Weight (N=8)
Pyrexia (General disorders) | 2 | 2 | 0
Fatigue (General disorders) | 0 | 2 | 1
Sepsis (Infections and infestations) | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypertension (Vascular disorders) | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/55/NCT03394755/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-09): https://cdn.clinicaltrials.gov/large-docs/55/NCT03394755/SAP_001.pdf